CLINICAL TRIAL: NCT02996019
Title: A Randomized, Open-Label, 2-Part, 2-Arm, Parallel-Group, Single-Dose, Multi-Center Study in Healthy Subjects to Investigate the Comparability of Pharmacokinetics of Etrolizumab Administered Subcutaneously by a Prefilled Syringe With Needle Safety Device or an Auto-Injector
Brief Title: A Study to Compare Pharmacokinetics (PK) of Etrolizumab Administered Subcutaneously by a Prefilled Syringe With Needle Safety Device (PFS-NSD) or an Auto-injector (AI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GX29504
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — etrolizumab

ARMS (4):
- Part 1: Etrolizumab AI (Experimental): Participants will receive a single dose of etrolizumab via subcutaneous (SC) injection using the AI on Day 1.
  Interventions: Drug: Etrolizumab; Device: Auto-Injector (AI)
- Part 1: Etrolizumab PFS-NSD (Active Comparator): Participants will receive a single dose of etrolizumab via SC injection using the PFS-NSD on Day 1.
  Interventions: Drug: Etrolizumab; Device: Prefilled Syringe With Needle Safety Device (PFS-NSD)
- Part 2: Etrolizumab AI (Experimental): Participants will receive a single dose of etrolizumab via SC injection using the AI on Day 1.
  Interventions: Drug: Etrolizumab; Device: Auto-Injector (AI)
- Part 2: Etrolizumab PFS-NSD (Active Comparator): Participants will receive a single dose of etrolizumab via SC injection using the PFS-NSD on Day 1.
  Interventions: Drug: Etrolizumab; Device: Prefilled Syringe With Needle Safety Device (PFS-NSD)

INTERVENTIONS:
Drug: Etrolizumab — Etrolizumab will be administered at a dose of 105 milligrams (mg).
  Other Names: RO5490261
Device: Auto-Injector (AI) — The pre-filled AI will be used to administer etrolizumab.
  Arms: Part 1: Etrolizumab AI; Part 2: Etrolizumab AI
Device: Prefilled Syringe With Needle Safety Device (PFS-NSD) — The PFS-NSD will be used to administer etrolizumab.
  Arms: Part 1: Etrolizumab PFS-NSD; Part 2: Etrolizumab PFS-NSD

SUMMARY:
This is a randomized, 2-part, 2-arm, open-label, parallel-group, multi-center study to compare the PK of etrolizumab administered subcutaneously by an AI (test device) or a PFS-NSD (reference device) in healthy participants. The study will comprise a pilot cohort (Part 1) to estimate the geometric mean ratio (GMR) and variability of the maximum observed concentration (Cmax) and area under the concentration-time curve (AUC) to confirm or determine the sample size for the pivotal cohort (Part 2). The pivotal cohort will demonstrate exposure comparability of Cmax, AUC from Hour 0 to the last measurable concentration (AUClast), and AUC from Hour 0 to extrapolated infinite time (AUC0-inf), values for a single dose of etrolizumab administered subcutaneously either by the AI or the PFS-NSD.

ELIGIBILITY:
Inclusion Criteria:

* Within the body weight range of 60 to 100 kilograms, inclusive (for the pivotal cohort [Part 2] only)
* Within body mass index (BMI) range 18.0 to 30.0 kilograms per square meter (kg/m^2), inclusive
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), and vital signs
* Females will be non-pregnant, non-lactating, and either postmenopausal (at least 12 months of non-therapy-induced amenorrhea)/surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days prior to enrolment, or agree to remain abstinent/use a highly effective method of contraception for at least 24 weeks after study drug administration
* Males will either be sterile or agree to remain abstinent/use a highly effective method of contraception for at least 24 weeks after study drug administration. Male participants will refrain from sperm donation from Check-in (Day -1) until 24 weeks following study drug administration

Exclusion Criteria:

* Any prior treatment with etrolizumab or other anti-integrin agents (including natalizumab, vedolizumab, and efalizumab)
* Any prior treatment with anti-mucosal addressin cell adhesion molecule 1 (anti-MAdCAM-1) agents
* Any prior treatment with rituximab
* Received intravenous corticosteroids within 30 days prior to Screening
* Use of agents that deplete B or T cells (e.g., alemtuzumab, rituximab, or visilizumab) within 12 months prior to randomization
* Any prior immunosuppressive agents (including cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil)
* Chronic nonsteroidal anti-inflammatory drug (NSAID) use
* Use of any prescription medications/products within 14 days prior to Check in (Day -1)
* History of demyelinating disease
* Neurological conditions or diseases
* History of cancer
* History of alcoholism or drug addiction within less than (<) 1 year prior to Screening
* History of active or latent tuberculosis (TB), regardless of treatment history
* History of recurrent opportunistic infections and/or history of severe disseminated viral infections
* Positive for human immunodeficiency virus (HIV) antibody
* Any current or recent signs or symptoms of infection
* Pregnant or lactating
* Hospitalized within 4 weeks prior to and during Screening
* History of organ transplant
* Presence of skin rash at Screening or history of other skin disorders
* Tattoos, scars, chronic rashes, or sunburn in the area of the designated injection site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Cmax of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 1: AUClast of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 1: AUC0-inf of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 1: Ratio of AUClast to AUC0-inf (AUCR) of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: Cmax of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: AUClast of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: AUC0-inf of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)

SECONDARY OUTCOMES:
Part 1: Time to Maximum Observed Concentration (tmax) of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: tmax of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 1: Apparent Terminal Elimination Half-Life (t1/2) of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: t1/2 of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Part 2: AUCR of Etrolizumab | Predose (0 hours) and 6 hours postdose on Day 1, on Days 2, 4, 6, 8, 11, 15, 29, 43, 57, and at end of study (Day 71) or early discontinuation (up to Day 71)
Percentage of Participants With Adverse Events | Part 1 and 2: Baseline up to Day 71
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) Against Etrolizumab | Part 1 and 2: Baseline up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Covance Research Unit - Daytona, Daytona Beach, Florida
  - Covance Clinical Research Unit Inc.; Covance Gfi Research, Evansville, Indiana
  - Covance Research Unit - Dallas, Dallas, Texas
  - Covance Clinical Research Unit, Inc, Madison, Wisconsin

REFERENCES:
- [Derived] Zhang W, Tyrrell H, Ding HT, Pulley J, Boruvka A, Erickson R, Abouhossein M, Ravanello R, Tang MT. Comparable Pharmacokinetics, Safety, and Tolerability of Etrolizumab Administered by Prefilled Syringe or Autoinjector in a Randomized Trial in Healthy Volunteers. Adv Ther. 2021 May;38(5):2418-2434. doi: 10.1007/s12325-021-01661-6. Epub 2021 Mar 29. PMID 33778929